CLINICAL TRIAL: NCT06394973
Title: Efficacy and Safety Assessment of T4090 Ophthalmic Solution (Preservative-free Kinezodianone R HCl 0.2% or 0.3%) Versus Rhopressa® Ophthalmic Solution (Preserved Netarsudil 0.02%) in Patients With Open-angle Glaucoma or Ocular Hypertension
Brief Title: Efficacy and Safety Assessment of T4090 Ophthalmic Solution Versus Rhopressa® Ophthalmic Solution in Patients With Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT4090-201
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- T4090 0.2% (Experimental)
  Interventions: Drug: T4090 0.2%
- T4090 0.3% (Experimental)
  Interventions: Drug: T4090 0.3%
- Rhopressa® (Active Comparator)
  Interventions: Drug: Rhopressa®

INTERVENTIONS:
Drug: T4090 0.2% — 1 drop in the conjunctival cul-de-sac of each eye once daily at 8:00 PM (±1 hour) from Day 1 to the day before the End of treatment visit (Visit #5 - Week 7).
  Arms: T4090 0.2%
Drug: T4090 0.3% — 1 drop in the conjunctival cul-de-sac of each eye once daily at 8:00 PM (±1 hour) from Day 1 to the day before the End of treatment visit (Visit #5 - Week 7).
  Arms: T4090 0.3%
Drug: Rhopressa® — 1 drop in the conjunctival cul-de-sac of each eye once daily at 8:00 PM (±1 hour) from Day 1 to the day before the End of treatment visit (Visit #5 - Week 7).
  Arms: Rhopressa®

SUMMARY:
The main purpose is to compare the ocular hypotensive efficacy and safety of two concentrations of T4090 (Kinezodianone R HCl 0.2% and 0.3%) ophthalmic solution with Rhopressa® ophthalmic solution

ELIGIBILITY:
Main Inclusion Criteria:

* Patient (male or female) ≥18 years old
* Patient with Open Angle Glaucoma or Ocular Hypertension in both eyes
* Informed consent dated and signed.

Main Exclusion Criteria:

* Secondary Open Agle Glaucoma (ex. Pseudoexfoliation, Pigmentary glaucoma)
* Advanced stage of glaucoma
* History of ocular trauma, eye infection, or/and ocular clinically significant inflammation within the 6 previous months.
* Known or suspected hypersensitivity to one of the components of the IMPs or other product used in the clinical study
* Pregnancy (confirmed with a positive urine pregnancy test) or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Arizona Advanced Eye Research Institute, Glendale, Arizona
  - Global Research Management, Inc., Glendale, California
  - United Medical Research Institute, Inglewood, California
  - Eye Research Foundation, Newport Beach, California
  - Visionary Research Institute, Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Sacramento Eye Consultants, A Medical Corporation, Sacramento, California
  - Wolstan and Goldberg Eye Associates, Torrance, California
  - Segal Drug Trials, Inc, Delray Beach, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Shettle Eye Research, Inc., Largo, Florida
  - Mild Florida Eye Center, Mt. Dora, Florida
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Alterman, Modi and Wolter Ophthalmic Surgeons, Poughkeepsie, New York
  - James D. Branch, MD, Winston-Salem, North Carolina
  - Total Eye Care, PA, Memphis, Tennessee
  - Keystone Research, Austin, Texas
  - Glaucoma Associates of Texas, Dallas, Texas
  - Houston Eye Associates, Houston, Texas
  - DCT-Shah Research, LLC sba Discovery Clinical Trials, Mission, Texas
  - Emerson Clinical Research Institute, Falls Church, Virginia
  - Piedmont Eye Center, Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 161 patients randomized and 159 patients treated. 2 Patients did not receive a treatment due to randomization error in IRT.
Groups:
- T4090 0.2%: Preservative-free Kinezodianone R HCl 0.2%, ophthalmic solution.
- T4090 0.3%: Preservative-free Kinezodianone R HCl 0.3%, ophthalmic solution.
- Rhopressa®: Preserved netarsudil 0.02%, ophthalmic solution.
Period: Overall Study
Arm/Group | T4090 0.2% | T4090 0.3% | Rhopressa®
Started (Assignement was made at participant level, meaning both eyes were treated with the same intervention.) | 53 | 53 | 53
Completed | 48 | 48 | 49
Not Completed | 5 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T4090 0.2% | T4090 0.3% | Rhopressa® | Total
Number analyzed (Participants) | 53 | 53 | 53 | 159
Age, Categorical [Count of Participants; unit: Participants] — Age by class
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 9 | 15 | 12 | 36
    >=65 years | 44 | 38 | 41 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at screening
  years | 71.4 (9.37) | 69.2 (9.45) | 70.3 (10.15) | 70.3 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 31 | 26 | 80
  Male | 30 | 22 | 27 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 11 | 11 | 35
  Not Hispanic or Latino | 40 | 42 | 42 | 124
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 9 | 12 | 9 | 30
  White | 42 | 40 | 42 | 124
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 53 | 53 | 53 | 159

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal IOP
Description: IOP measurement with calibrated Goldmann applanation tonometer in each eye at three time points (8:00 AM; 10:00 AM; 4:00 PM) by the Investigator.
  Mean diurnal is calculated from these three timepoints.
Time Frame: The primary efficacy endpoint is the change from baseline (D1) at Week 7 in the mean diurnal IOP in the study eye.
Population: Primary estimand - Full Set Analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | T4090 0.2% | T4090 0.3% | Rhopressa®
Number analyzed (Participants) | 45 | 42 | 47
mmHg | -5.07 (2.75) | -4.73 (2.94) | -4.6 (3.06)
Statistical Analysis 1: Comparison: T4090 0.2% vs Rhopressa®; Test type: Other; p = 0.376, Mixed Models Analysis; Mean Difference (Final Values) = -0.49
Statistical Analysis 2: Comparison: T4090 0.3% vs Rhopressa®; Test type: Other; p = 0.518, Mixed Models Analysis; Mean Difference (Final Values) = -0.36

ADVERSE EVENTS:
Time Frame: Adverse events were collected from informed consent signature (Visit #1) until the final study visit (Visit #5), up to 53 days.
Arm/Group | T4090 0.2% | T4090 0.3% | Rhopressa®
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 1/53
Other Adverse Events (participants affected / at risk) | 46/53 | 46/53 | 36/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T4090 0.2% (N=53) | T4090 0.3% (N=53) | Rhopressa® (N=53)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T4090 0.2% (N=53) | T4090 0.3% (N=53) | Rhopressa® (N=53)
Abnormal sensation in eye (Eye disorders) | 1 | 4 | 2
Blepharitis (Eye disorders) | 1 | 2 | 3
Conjunctival haemorrhage (Eye disorders) | 2 | 3 | 1
Conjunctival hyperaemia (Eye disorders) | 35 | 25 | 21
Corneal endothelial cell loss (Eye disorders) | 6 | 8 | 2
Corneal endothelial disorder (Eye disorders) | 19 | 16 | 11
Eye irritation (Eye disorders) | 2 | 5 | 2
Eye pain (Eye disorders) | 2 | 3 | 1
Eye pruritus (Eye disorders) | 5 | 6 | 4
Foreign body sensation in eyes (Eye disorders) | 3 | 5 | 3
Lacrimation increased (Eye disorders) | 5 | 8 | 6
Ocular hyperaemia (Eye disorders) | 5 | 9 | 7
Vision blurred (Eye disorders) | 7 | 7 | 4
Instillation site erythema (General disorders) | 5 | 8 | 2
Instillation site irritation (General disorders) | 4 | 8 | 10
Instillation site lacrimation (General disorders) | 5 | 2 | 1
Conjunctival staining (Investigations) | 3 | 1 | 1
Corneal pachymetry (Investigations) | 6 | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT06394973/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT06394973/SAP_001.pdf